CLINICAL TRIAL: NCT03894293
Title: Correlations Among Functional Performance, Muscle Strength and Weaning Rate in Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-02-006C
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Failure; Functional Performance; Physical Therapy
Keywords: functional performance; respiratory failure; weaning; mechanical ventilator; physical therapy; cardiopulmonary physical therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ventilator group: It's a observational study. Participants entry the Respiratory Care Center and are evaluated. If the participant meet the inclusion criteria, the first assessments will be collected. After the weaning training, the second assessment will be collected before the the endotracheal tube is removed.

SUMMARY:
To assess the correlations among the physical functional performance, muscle strength, respiratory muscle strength and the ventilator weaning rate.

DETAILED DESCRIPTION:
To assess the correlations among the physical functional performance, muscle strength, respiratory muscle strength and the ventilator weaning rate. Investigators use the DEMMI and FSS-ICU to evaluation the physical functional performance. And MRC score and hand dynamometer to record the muscle strength. The weaning parameters include Pi, PE, RSI,minute ventilation, tidal volume and cuff leak will be recorded. After the participant enters the Respiration Care Center, Doctor and physical therapist evaluate the consciousness and meet the inclusion criteria and the participant will received the first evaluation. The second evaluation will be held before the ventilator weaning timing.

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure with mechanical ventilator use
* 48 hours after transferring to respiratory care center
* consciousness clear and can obey orders
* vital signs stable

Exclusion Criteria:

* conscious disturbance
* neuromuscular disease
* stroke
* fracture
* patho fracture
* BMI>45

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory failure with mechanical ventilator user
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-02-19 (Estimated); Study Completion 2020-02-19 (Estimated)

PRIMARY OUTCOMES:
correlations between the Change from Baseline 'de Morton Mobility Index (DEMMI)' to the timing before weaning and the ventilator days | from baselineto the timing before weaning
  Correlations between the Functional physical performance and the ventilator days.It contains 5 items including bed skill, chair skills, static balance, walking and dynamic balance. The scores of 'bed', 'chair', 'static balance', 'walking' range from 0 to 4. And the score of 'dynamic balance' range from o to 3. The sum of 5 items is total raw score. Total Raw score is 0 to 19. And raw score can be converted to DEMMI score, ranging from 0 to 100. Higher values represent better mobility performance.
Correlations between the Change from Baseline 'Functional Status Score for the ICU (FSS-ICU)' to the timing before weaning and the ventilator days | from baselineto the timing before weaning
  Correlations between the Functional physical performance and the ventilator days.It contains 5 items including rolling, supine-to-sit, unsupported sit, sit-to-stand and ambulation. The scores of 5 items range from 0 to 7. 0 means unable to perform; 1 means total assistance; 2 means maximum assistance; 3 means moderate assistance; 4means minimal assistance; 5 means supervision; 6 means moderate independence and 7 means complete independence. The total score ranges from 0 to 35. Higher values represent better functional performance.

SECONDARY OUTCOMES:
Correlations between the Change from Baseline 'grip - hand strength' to the timing before weaning and ventilator days | from baselineto the timing before weaning
  Correlations between the hand strength and ventilator days. The measurement unit is kilogram(kg). The measurement tool is Jamar® Plus+ Digital Hand Dynamometer. Participant is required to use the best effort to squeeze 15 seconds and repeat 3 times. Resting time is 30 seconds. Investigators record the data and calculate the average data.
Correlation between the Change from Baseline 'Medical Research Council (MRC) scale' to the timing before weaning and ventilator days | baseline, before weaning
  Muscle strength assessment. 'Medical Research Council (MRC) scale' is an assessment tool of limb muscle strength. Left and Right sides are all tested. The Upper limb muscle tests include 'shoulder abduction', 'elbow flexion' and 'wrist extension. The lower limb muscle tests include 'hip flexion', 'knee extension' and 'ankle dorsiflexion'. The grades range from 0 to 5. Grade 0 means 'no contraction visible or palpable'; Grade 1 means 'flick of contraction visible or palpable, although no limb movement'; Grade3 means 'movement with gravity eliminated over almost full range of motion'; Grade 4 means 'movement against moderate resistance over full range of motion'; Grade 5 means 'normal power'. The sum of 6 items are total strength score which ranges from 0 to 60. Higher value represents better muscle strength. If the sum is below 48 points, it represents critical illness.
Correlations between the Change from Baseline 'Maximal inspiration pressure(PI)' to the timing before weaning and ventilator days | from baselineto the timing before weaning
  Evaluate the inspiratory muscle strength.Instruct the participants exhale slowly and completely, and then try to breath in as hard as possible. The participants should maintain inspiratory pressure for at least 1.5 seconds and the largest negative pressure sustained for at least one second should be recorded. The unit is cm H2O. Higher value represent better inspiratory muscle strength.
Correlation between the Change from Baseline 'Maximal expiration pressure(PE)' to the timing before weaning and ventilator days | from baselineto the timing before weaning
  Evaluate the inspiratory muscle strength.Instruct the participants inhale slowly and completely, and then try to breath out as hard as possible. The participants should maintain expiratory pressure for at least 1.5 seconds and the largest positive pressure sustained for at least one second should be recorded. The unit is cm H2O. Higher value represent better expiratory muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor ED, Walsham J. Should we mobilise critically ill patients? A review. Crit Care Resusc. 2009 Dec;11(4):290-300. PMID 20001881
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703